CLINICAL TRIAL: NCT01618253
Title: Phase I Study of Radiation Therapy With Concurrent Sorafenib for Hepatocellular Carcinoma Not Responding to Transarterial Chemoembolization
Brief Title: Radiation Therapy With Sorafenib for TACE-Resistant Hepatocellular Carcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Closed due to poor accrual.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00017344
Record Dates: First submitted 2012-06-04; First posted 2012-06-13 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer; Hepatoma; Liver Cancer
Keywords: Transarterial Chemoembolization; TACE; Sorafenib Tosylate; Sorafenib; Nexavar; External Beam Radiation Therapy; Radiation Therapy; Radiotherapy; Radiation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Sorafenib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiation therapy with concurrent sorafenib (Experimental)
  Interventions: Drug: Sorafenib; Radiation: Conventional fractionation (2 Gy per day) external beam radiation therapy

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400 mg PO bid will be started two weeks prior to initiation of radiation therapy (RT) and continue until the end of protocol specified radiation dose.
  Other Names: Sorafenib Tosylate; Nexavar
Radiation: Conventional fractionation (2 Gy per day) external beam radiation therapy — Patients will be stratified by the maximum diameter of HCC in any plane (≤10 cm or >10 cm) based on post-TACE, contrast enhanced MRI or CT. If only 1 lesion is present, the maximum diameter of that lesion in any plane determines stratification. If >1 but ≤3 lesions are present, the sum of the maximum diameter in any plane of all the lesions determines stratification.
  The MTD will be determined utilizing a standard 3 + 3 dose escalation scheme (4 Gy increase per bin). For lesions ≤10 cm, the starting RT dose bin will be 42 Gy and escalate to a pre-determined maximum of 62 Gy if no DLT's are experienced. For lesions >10 cm, the starting RT dose bin will be 40 Gy and escalate to a pre-determined maximum of 52 Gy if no DLT's are experienced.
  Other Names: External Beam Radiation Therapy; Radiation Therapy; Radiotherapy

SUMMARY:
To determine the maximum tolerated radiation dose with concurrent sorafenib for unresectable hepatocellular carcinoma that has not responded to transarterial chemoembolization.

DETAILED DESCRIPTION:
In patients with unresectable hepatocellular carcinoma (HCC), transarterial chemoembolization (TACE) is first line therapy. Non-responders to TACE (i.e. stable or progressive disease) represent a poor prognosis population with limited options. Sorafenib is indicated for first line salvage therapy, however it only improves survival 2-3 months and just has a 2-3% response rate. Thus, sorafenib is merely a cytostatic agent that delays progression and does not cytoreduce disease.

Radiation therapy (RT) is a non-invasive treatment that can cytoreduce HCC with minimal morbidity using modern techniques. A meta-analysis and multiple retrospective series suggest TACE + RT improve survival when compared to TACE alone. Higher RT doses are similarly associated with increased survival due to improved local control. Paradoxically, some series suggest that RT can induce vascular endothelial growth factor (VEGF) expression which may stimulate HCC.

Pre-clinical data suggest that combining RT with concurrent sorafenib (a VEGF inhibitor) improves tumor control. However, clinical data is limited to case reports and safety has not been well characterized. Prior to determining if this combination can improve control of HCC in this poor prognosis population, the optimal radiation dose with concurrent sorafenib must be determined by a phase I dose escalation trial.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic or histologic diagnosis of hepatocellular carcinoma (HCC).
* Maximum of 3 HCC lesions within the liver.
* No evidence of lymphadenopathy or metastatic disease per either CT or PET.
* Prior transarterial chemo-embolization (TACE) at least 28 days prior to initiation of protocol therapy.
* Evidence of either progressive disease or stable disease following TACE.
* Child Pugh Class A (score 5-6) or B (score 7).
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1 (or Karnofsky ≥70%).
* Normal organ and marrow function (platelets >60,000/mc; hemoglobin ≥8.5 g/dL; international normalized ratio (INR) ≤2.3; albumin ≥2.8 g/dL; total bilirubin ≤3 mg/dL; aspartate aminotransferase (AST) / alanine aminotransferase (ALT) <5x upper limit of normal; creatinine ≤1.5x upper limit of normal).
* Negative human immunodeficiency virus serology.
* Negative pregnancy test for women of child bearing age.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Less than 800 cc of normal liver.
* Child Pugh Class B (score 8-9) or C (score 10-15).
* Acute/active hepatitis B infection.
* Prior systemic chemotherapy or abdominal radiation therapy.
* Portal venous (main, primary right, or primary left trunks) or inferior vena cava thrombosis.
* Prior malignancy within 5 years of enrollment except for non-melanoma skin cancer.
* Prior history of myocardial infarction, cerebrovascular accident, or esophageal variceal bleed in the last 6 months.
* Pre-existing heart failure with either a clinical classification of New York Heart Association Class III or IV or cardiac ejection fraction of <45%.
* Systolic blood pressure > 160 mmHg or diastolic pressure > 100 mmHg despite optimal medical management.
* Pulmonary hemorrhage or other serious bleeding event (grade 2+) within 4 weeks initiation of protocol therapy.
* Prior history of scleroderma or active systemic lupus erythematosus.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | From date of enrollment until 3 months after completion of treatment.
  Maximum tolerated dose (MTD) will be determined by dose limiting toxicity (DLT) that is observed in either the acute (during treatment) or subacute (up to 3 months after treatment) setting. Acute DLT will be defined by grade 3-5 hepatic, gastrointestinal, dermatologic, hematologic, or pulmonary toxicity per Common Toxicity Criteria for Adverse Effects (CTCAE), v4.0. Subacute DLT will be defined by radiation induced liver disease (RILD) or grade 3-5 gastrointestinal, hematologic, or pulmonary toxicity per CTCAE, v4.0.

SECONDARY OUTCOMES:
Radiographic Response | 1 & 3 months post-treatment.
  Evaluated by either contrast enhanced MRI (preferred) or CT.
Patterns of Failure | From date of enrollment until the date of first documented progression, last known folow-up, or date of death from any cause, whichever came first, assessed up to 10 years.
  Classified as local (in-field), regional (intrahepatic out-of-field), or distant (extrahepatic, which includes porta hepatic lymph nodes).
Progression Free Survival | From date of enrollment until the date of first documented progression, last known folow-up, or date of death from any cause, whichever came first, assessed up to 10 years.
  From date of enrollment until first local, regional, or distant failure following RT, last follow-up, or death from any cause.
Overall Survival | From date of enrollment until the date of last known folow-up or date of death from any cause, whichever came first, assessed up to 10 years.
  From date of enrollment until last follow-up or death.
Health Related Quality of Life | 1, 2, & 3 months post-treatment.
  FACT-Hep survey will be utilized to establish pre-treatment baseline and then compared to post-treatment evaluations at months 1, 2, and 3.

CONTACTS AND LOCATIONS:
Overall Officials: Beth A. Erickson-Wittmann, M.D., Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Chung YL, Jian JJ, Cheng SH, Tsai SY, Chuang VP, Soong T, Lin YM, Horng CF. Sublethal irradiation induces vascular endothelial growth factor and promotes growth of hepatoma cells: implications for radiotherapy of hepatocellular carcinoma. Clin Cancer Res. 2006 May 1;12(9):2706-15. doi: 10.1158/1078-0432.CCR-05-2721. PMID 16675562
- [Background] Plastaras JP, Kim SH, Liu YY, Dicker DT, Dorsey JF, McDonough J, Cerniglia G, Rajendran RR, Gupta A, Rustgi AK, Diehl JA, Smith CD, Flaherty KT, El-Deiry WS. Cell cycle dependent and schedule-dependent antitumor effects of sorafenib combined with radiation. Cancer Res. 2007 Oct 1;67(19):9443-54. doi: 10.1158/0008-5472.CAN-07-1473. PMID 17909054
- [Background] Ren ZG, Zhao JD, Gu K, Chen Z, Lin JH, Xu ZY, Hu WG, Zhou ZH, Liu LM, Jiang GL. Three-dimensional conformal radiation therapy and intensity-modulated radiation therapy combined with transcatheter arterial chemoembolization for locally advanced hepatocellular carcinoma: an irradiation dose escalation study. Int J Radiat Oncol Biol Phys. 2011 Feb 1;79(2):496-502. doi: 10.1016/j.ijrobp.2009.10.070. Epub 2010 Apr 24. PMID 20421145